CLINICAL TRIAL: NCT06849310
Title: Intervention Protocol: Evaluation of the Effectiveness of the Emotion Regulation Program for Adolescents
Brief Title: Emotional Management in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Merve Oral, Lecturer, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-14588481-605.99-101274183
Record Dates: First submitted 2025-02-08; First posted 2025-02-27 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Emotional Regulation; Examining the Emotion Regulation Effectiveness to be Given to Adolescents
Keywords: adolescence; emotion; regulation; school
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This study was planned as a randomized controlled trial. The 9th and 10th grades of two high schools with the same status in the capital of Türkiye will constitute the sample of the research. Students in one high school will form an intervention group of 40 people, and students in the other high school will form a control group of 40 people. The emotion management program will be applied to the intervention group, and after the program is completed, the control group will be given information about the subject from an ethical point of view and a program booklet. The 40 children in the initiative group will be divided into groups. There will be an average of 13-14 people in each group. A 4-week intervention program will be applied to each group, 50 minutes per week.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants who will receive emotion regulation training. (Experimental): This study was planned as a randomized controlled trial. The 9th and 10th grades of two high schools with the same status in the capital of Türkiye will constitute the sample of the research.Adolescents will be randomized as an intervention and control group after stratification according to the mean score of the scale, gender (girls/boys), and grades (9th and 10th grades). Letters will be given to the intervention and control groups. According to the coin toss method, the letter A will be given to the initiative group and the letter B will be given to the control group. Randomization will be performed by a statistician independent of the research using the www.randomizer.org site. Adolescents will not be informed that they will be an intervention or control group. Criteria for inclusion in the research; (a) continuing their education in the 9th-10th grade, (b) agreeing to participate in the study, (c) giving written consent to participate in the study by their parents, (d) stating t
  Interventions: Behavioral: Group that will receive emotional regulation training
- Participants who will receive no intervention (No Intervention): All forms will be administered to adolescents in the control group twice, before and after the program (except for the descriptive characteristic data form). After the study is completed, the control group will be given the same training and written material.

INTERVENTIONS:
Behavioral: Group that will receive emotional regulation training — The content of the program is based on the current literature (Dennison, 2024; Holmqvist Larsson et al., 2020; Kara & Yüksel, 2022; Kılıçarslan & Varol, 2023; Siegel & Brayson, 2021; Vafaei et al., 2021) for four weeks, once a week (average 50 minutes/week). The module on noticing emotions, which will be applied in the first week, is aimed at adolescents to think about and notice emotions. The content of the training will include determining the beliefs and effects of the group members about emotions, teaching the nature of all emotions and the function of adaptation, distinguishing between emotions and thoughts, teaching similar and opposite emotions, and situations that contribute to the positivity of the emotional state.
  Arms: Participants who will receive emotion regulation training.

SUMMARY:
This study aims to give information about the content of the school-based emotion regulation program study designed for adolescent children to develop their emotion regulation skills. The study is a randomized controlled trial with adolescents aged 14-16 years (9th and 10th grade). Two high schools were selected for the research in Ankara, Türkiye. A face-to-face formal training consisting of four modules of four weeks (50 min/week). Based on the Vibrational Energy Theory, the program will be applied to the intervention group to be selected by the randomization method. The training topics include recognizing and accepting emotions, directed thinking and process orientation, and acceptance and willingness (reinforcement module) modules. With this intervention, adolescents' emotion regulation skills and psychological well-being are expected to increase, and anxiety levels will decrease. The program to be implemented will contribute to the acquiring and developing emotion regulation skills that deal with processes such as awareness, control, management, and acceptance of emotions in adolescents.

Key Words: adolescence, emotion, regulation, school

ELIGIBILITY:
Inclusion Criteria:

* . Criteria for inclusion in the research;

  * continuing their education in the 9th-10th grade,
  * agreeing to participate in the study,
  * giving written consent to participate in the study by their parents,
  * stating that they can participate in the four-week program,
  * speaking Turkish.

Exclusion Criteria:

* The criteria for exclusion from the study were:

  * the student has a medically diagnosed mental problem that will prevent the student from following the program,
  * the student has a psychological medical diagnosis, and
  * he/she is receiving psychiatric medication or therapy.

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
The Regulation of Emotions Questionnaire- REQ | 1 mounth
  The Regulation of Emotions Questionnaire (REQ) was developed by Phillips and Power (2007) to determine adolescents' emotion regulation methods. The scale consists of a total of 18 items and 4 sub-dimensions, including 5 Likert types (1 = Never, 5 = Always). Lower dimensions are classified as internal functional emotion regulation (4 items), internal dysfunctional emotion regulation (5 items), extrinsic functional emotion regulation (4 items), and extrinsic dysfunctional emotion regulation (5 items). The scale does not give a total score, scoring is done on the basis of sub-dimensions. As the scores obtained from the sub-dimensions increase, the frequency of the adolescent's emotion regulation method increases according to that sub-dimension, and as the score decreases, the rate of using that method decreases. There are no items that are scored backward. The reliability coefficients for the original study were .72 for intrinsic functional emotion regulation, .76 for dysfunctional emoti
The State-Trait Anxiety Inventory (STAI) | 1 mounth
  This scale was developed in 1970 by Spielberger et al. to measure the level of State and Trait Anxiety. The scale is used to determine how the individual feels in a certain condition and in a certain area. The scale can be applied to individuals aged 14 and over. The scale consists of two separate sub-scales, 20 of which were developed to measure state and 20 of which were developed to measure trait anxiety, consisting of a total of 40 items of Likert type. In this study, the State Anxiety Scale will be used. The feelings or behaviors specified in the State Anxiety Scale items are answered by choosing one of the options: 1: none, 2: somewhat, 3: a lot, and 4: completely, depending on the severity of such experiences (Spielberg et al., 1971). There are two types of expressions in the scale. These are either inverted or direct statements. Inverted statements express positive emotions, while direct expressions express negative emotions. Scoring on the State Anxiety Scale varies between
The Stirling Children's Well-being Scale (SCWBS) | 1 mounth
  It is a 5-point Likert model developed by Liddle and Carter (2015) to measure the emotional and psychological well-being levels of children aged 8-15 and rated between "Never (1) and Always (5)" consisting of 12 question items. There is no inverse matter on the scale. The highest score that can be achieved on the scale is 60, while the lowest score is 12. High scores obtained from the scale indicate that children's emotional and psychological well-being levels are high. In the original study, the internal consistency reliability coefficient of the scale was found to be .85 (Liddle & Carter, 2015). The scale was adapted into Turkish by Akın et al. in 2016. It was applied to primary, secondary, and high school students between the ages of 9-16. In the confirmatory factor analysis conducted for the adaptation studies to Turkish, it was seen that the one-dimensional model was well adapted. The Cronbach-Alpha internal consistency coefficient calculated within the scope of this study was fo

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol Üniversity, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/